CLINICAL TRIAL: NCT00711477
Title: Naltrexone Sustained Release (SR) 32 mg and Bupropion Sustained Release (SR) 360 mg Combination Therapy in Functional Magnetic Resonance Imaging (fMRI) Changes in Overweight or Obese Subjects
Brief Title: A Study Using Functional Magnetic Resonance Imaging (fMRI) to Assess the Effects of Naltrexone SR/ Bupropion SR Therapy in Overweight or Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NB-431
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Obesity
Keywords: obesity; overweight; magnetic resonance imaging; naltrexone; bupropion
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NB32 (Experimental): Naltrexone SR 32 mg/bupropion SR 360 mg/day
  Interventions: Drug: Naltrexone SR 32 mg/bupropion SR 360 mg/day; Other: fMRI scan
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo; Other: fMRI scan

INTERVENTIONS:
Drug: Naltrexone SR 32 mg/bupropion SR 360 mg/day
  Arms: NB32
Drug: Placebo
  Arms: Placebo
Other: fMRI scan — fMRI to assess the effects of the drug/placebo on areas of the brain
  Other Names: functional magnetic resonance imaging to assess the effects of the drug/placebo on areas of the brain

SUMMARY:
The purpose of this study was to assess the effect of naltrexone SR/bupropion SR (NB) on brain function in response to food cues using functional magnetic resonance imaging in overweight or obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed, female subjects, 18 to 45 years of age
* Body mass index (BMI) ≥ 27 and ≤ 40 kg/m²
* Free from clinically significant illness or disease as determined by medical history and physical examination
* Able to provide proof of identity during the enrollment process
* In good general health, without clinically significant medical history, physical examination findings or laboratory results
* Laboratory values obtained within 30 days of study entry within normal range for healthy volunteers.
* Normal urinalysis on initial screening day defined as: negative glucose, negative or trace protein, and negative or trace hemoglobin
* Normotensive (systolic ≤140 mm Hg, diastolic ≤90 mm hg)
* On no concomitant medications with the exception of oral contraceptives, vitamins, and over the counter pain, indigestion or allergy medication
* All women of child bearing potential must be non-lactating, must have a negative STAT pregnancy test, and agree to use effective contraception methods throughout study period and for 30 days after discontinuation of study drug. The following are considered effective methods of contraception: Combination or progestin-only birth control pills (oral contraceptives), vaginal contraceptive rings, contraceptive patches, Depo Provera, intrauterine devices, barrier methods with spermicide (condom/foam, diaphragm/ spermicide), abstinence. (Subjects who have had a tubal ligation, hysterectomy or are post-menopausal for 2 years are considered NOT to be of child bearing potential)
* For women not using hormonal methods of contraception, should be in the follicular phase of the menstrual cycle at the baseline visit.
* Non-smoker and no use of tobacco or nicotine products for at least 6 months prior to baseline. On screening and study days, we will test the subjects' urine for presence of nicotinine/cotinine (STAT) test as confirmatory evidence of being a non-smoker in addition to their self-report. A Tobacco Questionnaire and Breath CO will also be administered for eligibility on the day of screening for confirmation purposes.
* No clinically significant abnormality on ECG, baseline QTc <470
* Able to comply with all required study procedures
* Available for follow up for the duration of the study
* Willing and able to give written informed consent

Exclusion Criteria:

* Obesity of known endocrine or genetic origin (e.g., untreated hypothyroidism, Cushing's syndrome, Prader Willi Syndrome, established Polycystic Ovary Syndrome)
* Inability to participate in fMRI scanning sessions
* History of occupational exposure to metal flakes in their bodies or eyes.
* History of known indwelling ferromagnetic metals or fragments.
* History of acute or chronic illness that requires medical therapy including active gastrointestinal conditions that might interfere with drug absorption
* History or presence of hepatic, renal, cardiovascular or gastrointestinal diseases
* Type I or Type II diabetes mellitus requiring pharmacotherapy
* Active malignancy or history of malignancy (other than non-melanoma skin cancer or surgically cured cervical cancer) within 5 years of enrollment
* Serious psychiatric illness, including lifetime history of psychiatric hospitalization, suicide attempt, bipolar disorder, schizophrenia or other psychosis, bulimia, or anorexia nervosa; current serious personality disorder, (e.g. borderline or antisocial), major depressive disorder within the previous two years, suicidal ideation or need for psychiatric treatment in the previous 6 months.
* In need of medications for the treatment of a psychiatric disorder within the previous 6 months prior to randomization.
* IDS-SR total score >25 or scores >1 in items 5 (sadness), 6 (irritability), 7 (anxiety/tension) or 18 (suicidality)
* History of alcohol or drug abuse, current or within 2 years
* Unable to abstain from caffeinated product consumption for at least 48 hours
* History of surgical intervention for obesity
* Use of drugs, herbs, or dietary supplements believed to significantly affect body weight or participation in a weight loss management program within one month prior to randomization.
* History of hypersensitivity to bupropion or naltrexone
* History of seizure disorder or predisposition to seizures (e.g., history of cerebrovascular accident, brain surgery, head trauma with ≥5 minutes loss of consciousness, concussion symptoms lasting ≥ 15 minutes, skull fracture, subdural hematoma, or febrile seizures) or need for therapy with anticonvulsant medication.
* History of treatment with bupropion or naltrexone within 12 months
* Positive urine drug screen - STAT test performed on each day of study.
* Pregnant or breast-feeding
* Planned surgical procedure or trip that can impact the conduct of the study
* Use of investigational drug, device or procedure within 30 days
* Any condition which in the opinion of the investigator makes the subject unsuitable for inclusion in this study
* Participation in any previous clinical trial sponsored by Orexigen Therapeutics.
* Study personnel, sponsor representatives and their immediate families.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gene-Jack Wang, MD, Principal Investigator — Brookhaven National Laboratory
Locations (1):
- Brookhaven National Laboratory Medical Department, Upton, New York, United States

REFERENCES:
- [Background] Wang GJ, Tomasi D, Volkow ND, Wang R, Telang F, Caparelli EC, Dunayevich E. Effect of combined naltrexone and bupropion therapy on the brain's reactivity to food cues. Int J Obes (Lond). 2014 May;38(5):682-8. doi: 10.1038/ijo.2013.145. Epub 2013 Aug 8. PMID 23924756

RESULTS

PARTICIPANT FLOW:
Groups:
- NB32: Naltrexone SR 32 mg/day plus bupropion SR 360 mg/day
  fMRI scan: fMRI to assess the effects of the drug/placebo on areas of the brain
Period: Overall Study
Arm/Group | NB32 | Placebo
Started | 23 | 23
Completed | 20 | 20
Not Completed | 3 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Noncompliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | NB32 | Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.96 (7.68) | 30.39 (8.46) | 30.67 (7.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 8 | 20
  White | 3 | 8 | 11
  Other | 7 | 5 | 12
  Unknown or Not Reported | 0 | 1 | 1
Weight [Mean (Standard Deviation); unit: kg] | 87.70 (15.83) | 89.59 (13.34) | 88.64 (14.50)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.96 (4.30) | 31.80 (3.10) | 32.38 (3.75)

OUTCOME MEASURES:

1. Primary Outcome: Response to Food Related Cues Using Functional Magnetic Resonance Imaging - Superior Frontal
Description: Assessment of differences in brain activation in response to food cues before and after 4 weeks of treatment in subjects receiving NB or placebo.
Time Frame: Baseline, 4 weeks
Population: ITT (Intent-to-Treat): Included all subjects who were randomized, had a baseline measurement, and had at least one post-baseline fMRI measurement during the defined treatment phase.
Measure: Mean (90% Confidence Interval); unit: percent activation
Arm/Group | Placebo | NB32
Number analyzed (Participants) | 20 | 20
percent activation | -0.35 [-0.48 to -0.22] | 0.34 [0.21 to 0.47]
Statistical Analysis 1: Comparison: Placebo vs NB32; Test type: Superiority or Other; Mean Difference (Final Values) = 0.70, 90% CI 2-sided [0.50 to 0.90]

2. Secondary Outcome: Percent Change in Body Weight
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of body weight
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 20 | 20
percentage of body weight | -0.99 (0.44) | -0.43 (0.44)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.380, ANCOVA; Type III sums of squares from ANCOVA model: Treatment and Baseline; Mean Difference (Net) = -0.56, 95% CI 2-sided [-1.83 to 0.72]

3. Secondary Outcome: Dutch Eating Behavior Questionnaire - Change in Restrained Eating Subscale Score
Description: The Dutch Eating Behavior Questionnaire is a 33-item self-report measure designed to assess the type of eating behavior and is organized into 3 subscales (emotional eating, externally-induced eating, and restrained eating). Subjects rated the frequency of their eating behaviors using a 5-point scale, where 1=never, 2=seldom, 3=sometimes, 4=often, and 5=very often. The Restrained Eating subscale consisted of 10 items and the scores ranged from 10 (worse outcome) to 50 (better outcome).
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | 1.47 (0.86) | 1.87 (0.86)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.744, ANCOVA; Type III sums of squares from ANCOVA model: Treatment and Baseline; Mean Difference (Net) = -0.40, 95% CI 2-sided [-2.87 to 2.07]

4. Secondary Outcome: Dutch Eating Behavior Questionnaire - Change in Emotional Eating A Subscale Score
Description: The Dutch Eating Behavior Questionnaire is a 33-item self-report measure designed to assess the type of eating behavior and is organized into 3 subscales (emotional eating, externally-induced eating, and restrained eating). Subjects rated the frequency of their eating behaviors using a 5-point scale, where 1=never, 2=seldom, 3=sometimes, 4=often, and 5=very often. The Emotional Eating A subscale (clearly labeled emotions) consisted of 9 items and the scores ranged from 9 (better outcome) to 45 (worse outcome).
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -1.16 (0.77) | 0.48 (0.77)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.139, ANCOVA; Type III sums of squares from ANCOVA model: Treatment and Baseline; Mean Difference (Net) = -1.64, 95% CI 2-sided [-3.84 to 0.56]

5. Secondary Outcome: Dutch Eating Behavior Questionnaire - Change in Emotional Eating B Subscale Score
Description: The Dutch Eating Behavior Questionnaire is a 33-item self-report measure designed to assess the type of eating behavior and is organized into 3 subscales (emotional eating, externally-induced eating, and restrained eating). Subjects rated the frequency of their eating behaviors using a 5-point scale, where 1=never, 2=seldom, 3=sometimes, 4=often, and 5=very often. The Emotional Eating B subscale (diffuse emotions) consisted of 4 items and the scores ranged from 4 (better outcome) to 20 (worse outcome).
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -0.90 (0.55) | 0.45 (0.55)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.094, ANCOVA; Type III sums of squares from ANCOVA model: Treatment and Baseline; Mean Difference (Net) = -1.36, 95% CI 2-sided [-2.96 to 0.24]

6. Secondary Outcome: Dutch Eating Behavior Questionnaire - Change in External Eating Subscale Score
Description: The Dutch Eating Behavior Questionnaire is a 33-item self-report measure designed to assess the type of eating behavior and is organized into 3 subscales (emotional eating, externally-induced eating, and restrained eating). Subjects rated the frequency of their eating behaviors using a 5-point scale where 1=never, 2=seldom, 3=sometimes, 4=often, and 5=very often. The External Eating subscale consisted of 10 items and the scores ranged from 10 (better outcome) to 50 (worse outcome).
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -2.64 (1.03) | -0.16 (1.03)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.102, ANCOVA; Type III sums of squares from ANCOVA model: Treatment and Baseline; Mean Difference (Net) = -2.48, 95% CI 2-sided [-5.48 to 0.51]

7. Secondary Outcome: Change in Question 19 From 21-Item COE (Control of Eating) Questionnaire
Description: Question 19: Generally, how difficult has it been to control your eating? Scoring: 0=not at all difficult; 100=extremely difficult
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | -13.55 (4.67) | -4.14 (4.41)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.160, ANCOVA; Type III sums of squares from ANCOVA model: Treatment and Baseline; Mean Difference (Net) = -9.40, 95% CI [-22.7 to 3.89]

8. Primary Outcome: Response to Food Related Cues Using Functional Magnetic Resonance Imaging - Anterior Cingulate
Description: as for outcome 1
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: percent activation
Arm/Group | Placebo | NB32
Number analyzed (Participants) | 20 | 20
percent activation | -0.42 [-0.52 to -0.32] | 0.16 [0.04 to 0.28]
Statistical Analysis 1: Comparison: Placebo vs NB32; Test type: Superiority or Other; Mean Difference (Final Values) = 0.60, 90% CI 2-sided [0.40 to 0.80]

9. Primary Outcome: Response to Food Related Cues Using Functional Magnetic Resonance Imaging - Hippocampal Region 1
Description: as for outcome 1
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: percent activation
Arm/Group | Placebo | NB32
Number analyzed (Participants) | 20 | 20
percent activation | -0.16 [-0.32 to 0.00] | 0.60 [0.40 to 0.80]
Statistical Analysis 1: Comparison: Placebo vs NB32; Test type: Superiority or Other; Median Difference (Final Values) = 0.75, 90% CI 2-sided [0.50 to 1.00]

10. Primary Outcome: Response to Food Related Cues Using Functional Magnetic Resonance Imaging - Hippocampal Region 2
Description: as for outcome 1
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: percent activation
Arm/Group | Placebo | NB32
Number analyzed (Participants) | 20 | 20
percent activation | -0.79 [-0.99 to -0.59] | 0.21 [0.01 to 0.41]
Statistical Analysis 1: Comparison: Placebo vs NB32; Test type: Superiority or Other; Mean Difference (Final Values) = 0.99, 90% CI 2-sided [0.74 to 1.24]

11. Primary Outcome: Response to Food Related Cues Using Functional Magnetic Resonance Imaging - Superior Parietal
Description: as for outcome 1
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: percent activation
Arm/Group | Placebo | NB32
Number analyzed (Participants) | 20 | 20
percent activation | -0.56 [-0.87 to -0.25] | 0.74 [0.34 to 1.04]
Statistical Analysis 1: Comparison: Placebo vs NB32; Test type: Superiority or Other; Mean Difference (Final Values) = 1.30, 90% CI 2-sided [0.95 to 1.65]

12. Primary Outcome: Response to Food Related Cues Using Functional Magnetic Resonance Imaging - Posterior Insula
Description: as for outcome 1
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: percent activation
Arm/Group | Placebo | NB32
Number analyzed (Participants) | 20 | 20
percent activation | -0.16 [-0.25 to -0.07] | 0.30 [0.20 to 0.40]
Statistical Analysis 1: Comparison: Placebo vs NB32; Test type: Superiority or Other; Mean Difference (Final Values) = 0.44, 90% CI 2-sided [0.31 to 0.57]

ADVERSE EVENTS:
Time Frame: baseline to week 4
Description: The safety analysis set (i.e., all randomized subjects with at least one tablet of study treatment administered and with at least one investigator contact/assessment at any time after the start of study treatment, regardless of whether they completed the study) included 45 subjects (placebo, N=22; NB32, N=23)
Groups:
- NB32: Naltrexone SR 32 mg/day plus bupropion SR 360 mg/day
  fMRI scan: fMRI to assess the effects of the drug/placebo on areas of the brain fMRI scan: fMRI to assess the effects of the drug/placebo on areas of the brain
Arm/Group | NB32 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 10/23 | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NB32 (N=23) | Placebo (N=22)
Nausea (Gastrointestinal disorders) | 5 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Feeling abnormal (General disorders) | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon completion or termination of the CRADA, a final report including a list of inventions must be prepared and delivered to the Dept. of Energy Office of Scientific and Technical Information. Each party must provide the other with up to 45 days to review any proposed publication associated with the CRADA results. Approval of the planned publication will not be unreasonably withheld.